CLINICAL TRIAL: NCT00650429
Title: Ziprasidone Intramuscular/Oral In The Treatment Of Acute Exacerbation Of Schizophrenia Or Schizoaffective Disorder: A Six-Week Open Administration Study
Brief Title: A Study of the Efficacy and Safety of Ziprasidone for the Treatment of Acute Exacerbation of Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281056
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — IM ziprasidone at an initial dose of 10 or 20 mg for the first 3 days; additional doses could be administered according to clinical need, with the maximum total daily IM dose of 40 mg. On Day 4, IM treatment was switched to oral (PO) treatment at an initial dose of 40 mg twice daily for the first 2 days; doses could be subsequently adjusted within the range of 40 to 80 mg twice daily. Total treatment duration was 6 weeks.
  Other Names: Geodon, Zeldox

SUMMARY:
This study was conducted to examine the efficacy and tolerability of ziprasidone intramuscular (IM), and to assess the effect of switching from IM to oral ziprasidone for the treatment of acute exacerbation of schizophrenia and schizoaffective disorder in a Latin American population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder.
* Inpatients with acute exacerbation of psychotic symptoms.
* Patients with a minimum score of 40 on the BPRS scale (1-7).

Exclusion Criteria:

* Concurrent treatment with antipsychotic agents at study drug initiation (within 12 hours prior to study drug initiation); for depot agents a period of two weeks or one cycle, whichever is the longer, must occur between last administration and study drug initiation.
* Treatment with antidepressants or mood stabilizers within 7 days of start of ziprasidone.
* Patients currently receiving clozapine.
* Patients at immediate risk of committing harm to self or others.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-10; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in Brief Psychiatric Rating Scale (BPRS) total score | Screening, Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)

SECONDARY OUTCOMES:
Change from baseline to endpoint in Clinical Global Impressions-Severity (CGI-S) scale score | Screening, Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)
Change from baseline to endpoint in Clinical Global Impressions-Improvement (CGI-I) scale score | Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)
Simpson-Angus Scale (SAS) | Days 1 and 2 (IM), Day 4 (Switch), and Weeks 2 and 6 (PO)
Barnes Akathisia Scale (BAS) | Days 1 and 2 (IM), Day 4 (Switch), and Weeks 2 and 6 (PO)
Laboratory tests | Screening and Week 6
Electrocardiogram | Screening and Week 6
Adverse events | Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)
Abnormal Involuntary Movement Scale (AIMS) | Day 1 (IM), Day 4 (Switch), and Week 6 (PO)
Change from baseline to endpoint in Positive and Negative Syndrome Scale (PANSS) total score | Screening, Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)
Change from baseline to endpoint in Covi Anxiety Scale score | Screening, Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)
Change from baseline to endpoint in Positive PANSS subscale score | Screening, Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)
Change from baseline to endpoint in Negative PANSS subscale score | Screening, Days 1-3 (IM), Day 4 (Switch), Days 5-7 and Weeks 2, 4, and 6 (PO)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Mexico (4):
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, DF
  - Pfizer Investigational Site, Mexico City
  - Pfizer Investigational Site, Mexico D F

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281056&StudyName=A%20study%20of%20the%20efficacy%20and%20safety%20of%20ziprasidone%20for%20the%20treatment%20of%20acute%20exacerbation%20of%20schizophrenia%20or%20schizoaffective%20disorder